CLINICAL TRIAL: NCT06410807
Title: Development of Online Mind-body Training Programs for Adults With Subjective Cognitive Decline
Brief Title: Development of Web-Based Mind-Body Trainings for Adults With Subjective Concerns
Acronym: iMBT
Status: Completed | Type: Observational
Sponsor: Ohio State University (Other)
Responsible Party: Sponsor
Other Study IDs: 2023H0387
Record Dates: First submitted 2024-01-11; First posted 2024-05-13 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Aging; Focus Groups
Keywords: mindfulness-based stress reduction; cognitive function; mindfulness training; aging; subjective cognitive decline; focus groups; lifestyle education
MeSH Terms: interventions — Focus Groups

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adults with subjective cognitive decline: Five focus groups will be conducted with adults with subjective cognitive decline recruited in the greater Columbus, Ohio area.
  Interventions: Other: Focus groups

INTERVENTIONS:
Other: Focus groups — The present study consists of 5 focus groups over 3 waves to inform the development and refinement of internet-based mindfulness (iMBSR) and lifestyle education (iLifeEd) protocols for use in future clinical trials. 50% females and 50% minoritized participants will be recruited to ensure representation across sex and race. For all focus groups, adults (over the age of 50 years) who report SCD will be recruited. Specifically, the Everyday Cognition Questionnaire (E-Cog) will be administered to quantify informant-reported deficits in cognitive functioning.

SUMMARY:
The goal of this observational study is to develop online, self-paced mindfulness (iMBSR) and lifestyle education (iLifeEd) programs for adults with cognitive concerns. Participants will engage in focus groups to discuss healthy living, web-based behavioral interventions, intervention content/format and ideal outcomes after engaging in behavioral interventions that promote healthy living. Additionally, participants will provide feedback on the protocol and online platform for either iMBSR or iLifeEd. This feedback will be used to refine the iMBSR and iLifeEd protocols for future use in the randomized controlled trial portion of the parent project.

DETAILED DESCRIPTION:
Rising prevalence rates of Alzheimer's Disease (AD) have led to widespread interest in identifying individuals at-risk for AD and for developing interventions that delay or prevent the onset of AD. Growing evidence suggests that subjective cognitive decline (SCD)-characterized by perceived persistent declines in cognitive functioning compared to previously normal cognitive status-may be a preclinical stage of Alzheimer's Disease. Individuals with SCD can be identified by self-reported declines in cognitive functioning based on self-report questionnaires, such as the Everyday Cognition Questionnaire, yet also exhibit normal performance based on age, sex, and education corrected standardized cognitive measures. There is mounting evidence that mindfulness training, traditionally offered as an 8-week in-person MBSR program, improves cognitive functioning including in the investigators' pilot MBSR trial with healthy older adults. Further, recent evidence from adults over the age of 60 has linked trait mindfulness with lower accumulation of AD pathology, lower cognitive decline on measures of global cognition, sustained attention, and immediate and delayed memory. Together, this suggests that mindfulness training could be beneficial as a preventative training program in adults with SCD who have yet to show objective cognitive impairments. However, limited accessibility, time and schedule constraints, and travel logistics are among the greatest barriers for in-person MBSR programs. Internet-based mindfulness programs are a promising and cost-effective approach, but few studies have adapted MBSR for internet-delivery in an asynchronous format. Several internet-based interventions ideographically tailored for the target population, including acquired brain injury, fibromyalgia, and heart disease show promising support. The present study seeks to address the urgent need for the development of alternative training programs that provide theoretical promise for reducing age-related cognitive decline, demonstrate broad transfer effects to domains of cognitive functioning that directly impact everyday functioning, and facilitate the development of a mechanistic model with easily identifiable and separable mechanisms. The aim of the present study is to iteratively develop and refine internet-based MBSR (iMBSR) and internet-based lifestyle education (iLifeEd) protocols with a team of stakeholders (i.e., focus groups). Focus groups of adults with subjective cognitive decline will be recruited to iteratively develop and refine the platforms for the iMBSR and iLifeEd groups. The iMBSR program will be a promising platform to deliver evidence-based mindfulness meditation techniques. Additionally, the iLifeEd program that will match the iMBSR program in terms of format of delivery, duration of training, peer support, and homework assignment will be developed.

ELIGIBILITY:
Inclusion Criteria:

* 50 years of age or older
* Report subjective cognitive decline with normatively intact performance on cognitive testing
* Capable of attending the assessment and the majority of focus group sessions
* Fluent English speaker
* Corrected (near and far) visual acuity of 20/40 or better
* Adequate hearing for experimental purposes
* Absence of diagnosed terminal illness
* Absence of diagnosed neurological disorders
* No history of psychotic disorder or substance abuse disorder
* Absence of any psychiatric disorder that was 1) diagnosed by a psychologist or psychiatrist and 2) diagnosed within the past 2 years OR symptoms and/or treatment is ongoing
* Absence of medication use that significantly alters brain activity
* No history of diagnosed learning disability that would interfere with the completion of cognitive tasks
* No evidence of mild cognitive impairment (MCI) or dementia: >1 standard deviation (SD) below demographically adjusted normative mean on both measures of one domain OR >1 SD below demographically adjusted normative mean on at least one measure of all three domains OR inadequate self-reported performance of instrumental activities of daily living
* Able to engage in light stretching exercises with or without assistive devices
* No regular practice of meditation or yoga (defined as once or more per week) AND no previous participation in a structured mindfulness class such as MBSR
* Access to the internet

Exclusion Criteria:

* Not 50 years of age or older
* Does not report subjective cognitive decline AND/ OR does not perform in the normatively intact range on cognitive testing
* Any physical limitation or pragmatic limitation that prohibits attendance at assessment and focus group sessions
* No fluency in English
* Corrected (near or far) visual acuity worse than 20/40
* Self-reported hearing impairment that would affect their ability to hear the experimenter
* Diagnosis of terminal illness
* Presence of diagnosed neurological disorders
* History of psychotic disorder or substance abuse disorder diagnosed by a psychologist or psychiatrist
* Presence of any psychiatric disorder that was 1) diagnosed by a psychologist or psychiatrist and 2) diagnosed within the past 2 years OR symptoms/treatment is ongoing
* Medication use that significantly alters brain activity
* History of diagnosed learning disability that would interfere with completion of the cognitive tasks
* Evidence of MCI or dementia: >1 SD below demographically adjusted normative mean on both measures of one domain OR >1 SD below demographically adjusted normative mean on at least one measure of all three domains OR inadequate self-reported performance of instrumental activities of daily living
* Actual or perceived limitation that prohibits engaging in light stretching exercises with or without assistive devices
* Any regular practice of meditation or yoga (defined as once or more per week) OR previous participation in a structured mindfulness class such as MBSR
* No access to the internet

Min Age: 50 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adults aged 50 years and over in the greater Columbus area with subjective cognitive decline
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-05-02 (Actual); Study Completion 2025-05-02 (Actual)

PRIMARY OUTCOMES:
Qualitative themes derived from focus group discussions on healthy living, web-based behavioral interventions, intervention content/format and ideal outcomes after engaging in behavioral interventions that promote healthy living | Baseline
  Qualitative summary of perceptions and attitudes regarding healthy living, web-based lifestyle interventions, intervention content/format and ideal intervention outcomes
Qualitative themes derived from focus group discussions on perceptions of, attitudes toward, and feedback on initial intervention protocols | Baseline
  Qualitative summary of perceptions of, attitudes toward, and feedback on initial intervention protocols and how focus group feedback was incorporated into protocol development
Qualitative themes derived from focus group discussions on perceptions of, attitudes toward, and feedback on fully developed web-based interface of the iMBSR and iLifeEd programs | Baseline
  Qualitative summary of perceptions of, attitudes toward, and feedback on fully developed web-based interface of the iMBSR and iLifeEd programs

CONTACTS AND LOCATIONS:
Overall Officials: Ruchika Prakash, PhD, Principal Investigator — Ohio State University
Locations (1):
- Department of Psychology, The Ohio State University, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No